CLINICAL TRIAL: NCT02130765
Title: Substrate Targeted Ablation Using the FlexAbility™ Ablation Catheter System for the Reduction of Ventricular Tachycardia (STAR-VT) - G130132
Brief Title: Substrate Targeted Ablation Using the FlexAbility™ Ablation Catheter System for the Reduction of Ventricular Tachycardia
Acronym: STAR-VT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to low enrollment rate.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJM-CIP-0005
Record Dates: First submitted 2014-04-28; First posted 2014-05-05 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Monomorphic Ventricular Tachycardia
Keywords: Monomorphic Ventricular Tachycardia; Ischemic; Non-ischemic; Catheter Ablation
MeSH Terms: conditions — Ischemia | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Drug with ICD/CRT-D (No Intervention): Implantable cardioverter defibrillator (ICD) or Cardiac Resynchronization Therapy-Defibrillator (CRT-D) with routine drug therapy
- Cardiac catheter ablation with ICD/CRT-D (Active Comparator): Cardiac catheter ablation with ICD/CRT-D with routine drug therapy
  Interventions: Device: Cardiac catheter ablation with ICD/CRT-D

INTERVENTIONS:
Device: Cardiac catheter ablation with ICD/CRT-D — Cardiac ablation catheter system
  Arms: Cardiac catheter ablation with ICD/CRT-D

SUMMARY:
To demonstrate that scar-based ventricular tachycardia (VT) ablation using the FlexAbility™ ablation catheter system results in a superior clinical outcome compared to routine drug therapy in subjects with documented Monomorphic Ventricular Tachycardia [MMVT] (both ischemic and non-ischemic) while maintaining an acceptable safety profile.

DETAILED DESCRIPTION:
Approximately 50 centers in the United States (US) will participate in the study. Additional centers outside the US may be considered, as necessary. The anticipated enrollment duration is 48-60 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient is receiving a new St.Jude Medical (SJM) Implantable Cardioverter Defibrillator (ICD) or SJM Cardiac Resynchronization Therapy-Defibrillator (CRT-D) implant, which has study required programing capabilities and is appropriate for remote monitoring. Subjects who have received the ICD / CRT-D up to 90 days prior to enrollment are also eligible.
* Patient who has a high risk of ICD shock as shown by at least one documented Monomorphic VT (MMVT)** by one or more of the following:

Spontaneous MMVT or Inducible MMVT during electrophysiology (EP) Study or Inducible MMVT during Non-Invasive Programmed Stimulation (NIPS) Study

* 18 to 75 years of age
* Patient has been informed of the nature of the study and has agreed to its provisions and provided written informed consent approved by the Institutional Review Board.

  * Note Pleiomorphic ventricular tachycardia (VT) (multiple MMVT morphologies) is acceptable but polymorphic VT or ventricular fibrillation (VF) is not.

Exclusion Criteria:

* Any history of stroke
* S-T elevation myocardial infarction (MI) or previous cardiac surgery within 60 days prior to enrollment
* Patient is pregnant or nursing
* Patient has New York Heart Association (NYHA) class IV heart failure
* Patient has incessant ventricular tachycardia (VT) necessitating immediate treatment (Patients with Incessant VT have continuous sustained VTs that recur promptly despite repeated intervention for termination over several (≥3) hours)
* Patient has VT/VF thought to be from channelopathies
* Limited life expectancy (less than one year) according to Investigator
* Patient has current class IV angina
* Recent coronary artery bypass graft (CABG < 60 days) or percutaneous coronary intervention (PCI < 30 days)
* Patient is currently participating in another investigational drug or device study
* Patient is unable or unwilling to cooperate with the study procedures
* Known presence of intracardiac thrombi (i.e., positive Transesophageal Echocardiogram (TEE) for LA or LV clot). TEE is required for history of left atrium (LA) or left ventricle (LV) clot and recommended for history of atrial fibrillation (AF) with CHADS > 1
* Prosthetic mitral or aortic valve
* Mitral or aortic valvular heart disease requiring immediate surgical intervention
* Major contraindication to anticoagulation therapy or coagulation disorder
* Left Ventricular Ejection Fraction < 15%
* Patient has had a previous ablation procedure for ventricular tachycardia (VT), excluding remote (> 3 months) outflow tract tachycardia
* Patient has glomerular filtration rate (GFR) < 30 mL/min/1.73m2 within the past 3 months
* Patient has peripheral vascular disease that precludes LV access
* Patient has a premature ventricular contraction (PVC) or VT induced cardiomyopathy that is expected to resolve with ablation and will not require an ICD
* Patient has reversible cause of VT
* Use of left ventricular assist device (LVAD) or Tandem Heart devices (Impella and Balloon pumps are acceptable)
* There is a strong clinical reason to believe that, in the opinion of the investigator, the patient only has septal scar that is deep

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07-25 (Actual); Study Completion 2016-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation; Francis Marchlinski, MD, Principal Investigator — University of Pennsylvania
Locations (38):
- United States (30):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - USC University Hospital, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - University of California at San Diego (UCSD) Medical Center, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University Hospital, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Mid-America Cardiology Associates, Kansas City, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine - Barnes Jewish Hospital, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - New York University Hospital, New York, New York
  - New York University Langone Medical Center, New York, New York
  - Mt. Sinai Hospital, New York, New York
  - Staten Island University Hospital - North, Staten Island, New York
  - Sanger Clinic, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt Heart and Vascular Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - The Methodist Hospital, Houston, Texas
  - Memorial Hermann Hospital, The Woodlands, Texas
  - Intermountain Heart Rhythm Specialist, Murray, Utah
  - University of Washington Medical Center, Seattle, Washington
- Royale Adelaide Hospital, Adelaide, Australia
- France (4):
  - Hopital d'adulte de la Timone, Marseille, Alpes
  - CHU Trousseau, Chambray-lès-Tours, Centre-Val de Loire
  - Clinique Protestante, Lyon
  - Hôpital du Haut Lévêque, Pessac
- Ospedale San Raffaele, Milan, Lombardy, Italy
- United Kingdom (2):
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized Subjects-Ablation: Enrolled subjects who meet entry criteria and are randomized to the ablation group (Subjects to receive ablation therapy for ventricular tachycardia using the FlexAbility(TM) Ablation Catheter System in addition to routine drug therapy)
- Randomized Subjects- Control: Enrolled subjects who meet entry criteria and are randomized to the control group (Subjects to receive routine drug therapy)
- Registry Subjects: Enrolled subjects who do not meet entry criteria (specifically noninvasive programmed stimulation [NIPS] or electrophysiology [EP] study without monomorphic ventricular tachycardia [MMVT] and absence of spontaneous documented MMVT).
- Early Withdrawal Subjects: Subjects enrolled but withdrawn early from the study
Period: Overall Study
Arm/Group | Randomized Subjects-Ablation | Randomized Subjects- Control | Registry Subjects | Early Withdrawal Subjects
Started | 11 | 8 | 26 | 19
Completed | 7 | 8 | 26 | 19
Not Completed | 4 | 0 | 0 | 0
Not completed — Did not receive treatment | 4 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Subjects-Ablation | Randomized Subjects-Control | Registry Subjects | Early Withdrawal Subjects | Total
Number analyzed (Participants) | 11 | 8 | 26 | 19 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (5.9) | 61.3 (7.3) | 60.6 (10.8) | 58.4 (15.0) | 60.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 6 | 4 | 11
  Male | 10 | 8 | 20 | 15 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 5 | 4 | 10
  White | 9 | 6 | 21 | 13 | 49
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 21 | 17 | 50
  Italy | 1 | 0 | 5 | 1 | 7
  France | 4 | 2 | 0 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experienced an ICD Shock Event.
Description: Primary Effectiveness endpoint: Number reported is number of subjects who experienced an ICD shock event (including both appropriate and inappropriate) through 12 month follow up
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Registry Subjects: Enrolled subjects who do not meet entry criteria (specifically NIPS or EP Study without MMVT and absence of spontaneous documented MMVT).
Arm/Group | Randomized Subjects-Ablation | Randomized Subjects- Control | Registry Subjects | Early WIthdrawal Subjects
Number analyzed (Participants) | 7 | 8 | 26 | 19
Participants | 1 | 1 | 0 | NA — Primary effectiveness data not collected in early withdrawal subjects

2. Primary Outcome: Number of Subjects Who Experienced a Select Serious Adverse Event
Description: Primary Safety Endpoint: Number of subjects who experience a select serious adverse events within the 30 day follow up. Those events are anticipated, associated with catheter ablation, and are cardiovascular, pulmonary, or peripheral vascular in nature, as listed in the Primary Safety Events List.
Time Frame: 30 days
Population: 4 subjects randomized to treatment arm but did not receive ablation (not treated) and therefore excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Subjects-Ablation | Randomized Subjects- Control | Registry Subjects | Early Withdrawal Subjects
Number analyzed (Participants) | 7 | 8 | 26 | 19
Participants | 2 | NA — Primary safety events not measured in this arm because events required to be related to catheter ablation | NA — Primary safety events not measured in this arm because events required to be related to catheter ablation | NA — Primary safety events not measured in this arm because events required to be related to catheter ablation

3. Secondary Outcome: Number of Subjects That Had a Cardiovascular (CV) Hospitalizations or CV-related ER Visit
Description: Number of subjects that had a CV hospitalization or CV-related ER visit through 12 month follow up.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Subjects-Ablation | Randomized Subjects- Control | Registry Subjects | Early Withdrawal Subjects
Number analyzed (Participants) | 7 | 8 | 26 | 19
Participants | 3 | 1 | 2 | 0

ADVERSE EVENTS:
Description: Adverse event reporting occurred from the time of subject enrollment (time of signed informed consent) through subject's completion in the study, subject withdrawal, early study termination, or otherwise discontinuation from the study. Therefore adverse events are reported for all 64 enrolled subjects including all randomized subjects, registry subjects, and early withdrawal subjects for the duration of time each subject was enrolled in the study.
Groups:
- All Enrolled Subjects: All Enrolled Subjects
- Randomized Subjects- Ablation: Enrolled subjects who meet entry criteria and are randomized to the ablation group (Subjects to receive ablation therapy for ventricular tachycardia using the FlexAbility (TM) Ablation Catheter System in addition to routine drug therapy).
- Randomized Subjects-Control: Enrolled subjects who meet entry criteria and are randomized to the control group (Subjects to receive routine drug therapy).
Arm/Group | All Enrolled Subjects | Randomized Subjects- Ablation | Randomized Subjects-Control | Registry Subjects | Early Withdrawal Subjects
All-Cause Mortality (participants affected / at risk) | 1/64 | 0/11 | 0/8 | 1/26 | 0/19
Serious Adverse Events (participants affected / at risk) | 9/64 | 5/11 | 2/8 | 2/26 | 0/19
Other Adverse Events (participants affected / at risk) | 4/64 | 1/11 | 2/8 | 1/26 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=64) | Randomized Subjects- Ablation (N=11) | Randomized Subjects-Control (N=8) | Registry Subjects (N=26) | Early Withdrawal Subjects (N=19)
Acute Bacterial Endocarditis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated Thresholds (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral Arterial Occlusion (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature Ventricular Contraction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Regular Narrow QRS Tachycardia/Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sustained Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=64) | Randomized Subjects- Ablation (N=11) | Randomized Subjects-Control (N=8) | Registry Subjects (N=26) | Early Withdrawal Subjects (N=19)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erectile Dysfunction Symptoms (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Low enrollment rates resulted in early termination. Therefore the study did not reach the target number of participants needed to achieve target power and statistically reliable results, and statistical hypothesis testing was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No